CLINICAL TRIAL: NCT05970627
Title: Perioperative Chemotherapy Combined With PD-1 Inhibitor (Toripalimab) for Treatment of Epstein-Barr Virus-associated Locally Advanced Gastric or Esophagogastric Junction Adenocarcinoma: a Prospective, Multi-center, Phase II Study
Brief Title: Perioperative Chemotherapy Plus Toripalimab for Epstein-Barr Virus-associated Locally Advanced Gastric or Esophagogastric Junction Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yu jiren (Other)
Responsible Party: Sponsor-Investigator, Yu jiren, Director of gastrointestinal surgery department, First Affiliated Hospital of Zhejiang University
Organization: First Affiliated Hospital of Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20230033C-R1
Record Dates: First submitted 2023-07-25; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Adenocarcinoma of the Stomach; Adenocarcinoma of Esophagogastric Junction; Epstein-Barr Virus-Associated Gastric Carcinoma
Keywords: Gastric Adenocarcinoma; Esophagogastric Junction Adenocarcinoma; Perioperative Chemotherapy; Toripalimab; Epstein-Barr Virus-associated gastric cancer
MeSH Terms: interventions — toripalimab; Oxaliplatin; S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy+Toripalimab (Experimental): Toripalimab: 240 mg IV infusion on Day 1 of each 21 day cycle for 3 cycles prior to surgery and 3 cycles after surgery.
  Chemotherapy: SOX(S-1+Oxaliplatin) Oxaliplatin,administered as a 2-hour intravenous infusion (130mg/m2) S-1, orally twice daily for 2 weeks followed by a 7-day rest period. The dose of S-1 was 80 mg/day for body surface area less than 1.25 m2, 100 mg/day for body surface area greater than or equal to 1.25 to less than 1.5 m2, and 120 mg/day for body surface area greater than or equal to 1.5 m2 Chemotherapy will be repeated each 21 day for 3 cycles prior to surgery and 3 cycles after surgery.
  Interventions: Drug: Toripalimab; Drug: Oxaliplatin; Drug: S1

INTERVENTIONS:
Drug: Toripalimab — Perioperative Toripalimab, 240 mg IV infusion
Drug: Oxaliplatin — Oxaliplatin (130 mg/m2) infusion as perioperative chemotherapy
Drug: S1 — S-1 orally intake as perioperative chemotherapy

SUMMARY:
This study is a prospective, single arm, multi-center phase II clinical trial designed to evaluate the efficacy and safety of perioperative SOX combined with toripalimab in participants with Epstein-Barr Virus-associated locally advanced gastric or esophagogastric junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in the clinical study; fully understands and is informed of the study and has signed the Informed Consent Form (ICF).
2. Participants were ambulatory male or female. Age: ≥ 18 years and ≤ 80 years old.
3. Histopathologically confirmed gastric or esophagogastric junction adenocarcinoma.
4. Epstein-Barr Virus-associated Gastric or Esophagogastric Junction Adenocarcinoma, which was determined by in situ hybridization (ISH) test of endoscopic biopsy specimen.
5. cT2-4bN+/-, M0 according to the American Joint Committee on Cancer and Union for International Cancer Control (AJCC-UICC) TNM classification for carcinoma of the stomach (8th edition).
6. Participants had Eastern Cooperative Oncology Group (ECOG) performance status scores of 0-1 within 7 days before the first dose of study treatment.
7. Life expectancy ≥ 6 months.
8. Agreement of providing baseline and surgical specimens for biomarker analysis.
9. The functions of the vital organs meet requirements as follows (within 14 days before the first dose of study treatment, meanwhile, participants had not received treatment of recombinant human thrombopoietin or granulocyte stimulating factor):

1). Hematological function

* White blood cell count (WBC): 3.5 × 10^9/L ~12.0 × 10^9/L
* Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L
* Platelet count (PLT) ≥ 100 × 10^9/L
* Hemoglobin (Hb) ≥ 90g/L. 2). Hepatic function

  * Total bilirubin (TBIL) ≤ 1.5 × ULN (upper limit of normal); -Aspartate aminotransferase (AST) ≤ 2.5 × ULN;
  * Alanine aminotransferase (ALT) ≤ 2.5 × ULN;
  * Albumin (ALB) ≥ 30g/L. 3). Renal function
  * Creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance ≥ 60 ml/min for those with creatinine level > 1.5 × ULN.

    4). Coagulation function
  * International normalized ratio (INR) ≤ 1.5;
  * Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.

    10. Female participants of childbearing age must meet requirements: urine or serum pregnancy test must be negative within 7 days before the first dose of study treatment, and she must agree to use adequate contraception methods or keep abstinence (starting with the ICF is signed through 120 days after the last dose of toripalimab, or 180 days after the last dose of chemotherapy, whichever is longer, and should not be breastfeeding. Male participants must meet requirements: agree to use adequate contraception methods or keep abstinence (starting with the ICF is signed through 120 days after the last dose of toripalimab, or 180 days after the last dose of chemotherapy, whichever is longer).

Exclusion Criteria:

1. HER2-positive status defined as either IHC score of 3+ or IHC 2+ with amplification proven by fluorescent in situ hybridization (FISH) based on pretreatment endoscopic biopsies.
2. Prior systemic therapy for treatment of gastric cancer (surgery, chemotherapy, radiotherapy, targeted therapy or immunotherapy).
3. Previous or concurrent have other active malignant tumors within the past 5 years (except for basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, prostate cancer or cervical cancer or breast cancer in situ that has undergone curative therapy).
4. Participants with gastric outlet obstruction, or unable to oral take, or severe gastrointestinal bleeding.
5. Myocardial infarction within 6 months before the first dose of study treatment, uncontrolled angina, arrhythmia which need medical intervention (including but not limited to cardiac pacemaker), congestive heart failure (New York Heart Association (NYHA) class III or IV).
6. Existence of chronic diarrhea (watery diarrhea: ≥ 5 times per day).
7. Participants with active infection within 14 days before the first dose of study treatment which need medical intervention.
8. Participants with active tuberculosis.
9. Previous or concurrent diagnosed with interstitial lung disease by imaging or symptoms.
10. Any of the following test is positive: Human Immunodeficiency Virus (HIV) antibody, Hepatitis B surface Antigen (HBsAg), or Hepatitis C Virus (HCV) antibody.
11. Participants who need long-term systemic steroid therapy (> 10 mg/d prednisone equivalent) or any other form of immunosuppressive therapy within 14 days before the first dose of study treatment or during the study period.
12. Concurrent or previous have severe allergic reaction to any antibody based drugs.
13. Existence of any concurrent autoimmune disease, excepting participants with diabetes mellitus type I, hypothyroidism requiring only hormone replacement therapy.
14. Receive live vaccines within 28 days before the first dose of study treatment or during the study period, excepting inactivated viral vaccines for seasonal influenza.
15. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
16. Existence of systemic disease that is difficult to control despite treatment with several agents, for example, diabetes mellitus, hypertension, etc.
17. Existence of other serious physical or mental diseases or serious laboratory abnormalities that may increase the risk of participating in the study. Participants who were judged unsuitable as subjects of this trial by investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-28 (Estimated); Primary Completion 2026-07-28 (Estimated); Study Completion 2029-07-28 (Estimated)

PRIMARY OUTCOMES:
Rate of pathological complete responses (pCR) | From enrollment to surgery after pre-operative treatment (up to approximately 36 months)
  Percentage of patients with pCR referring to the total number of enrolled and eligible patients, as evaluated centrally by a reference pathologist.

SECONDARY OUTCOMES:
Overall survival | From randomization to the last follow-up or death from any cause (up to approximately 72 months)
  The duration of overall survival (OS) will be determined by measuring the time interval from enrollment to the end of follow up or death from any cause
Progression-free survival | From randomization to the last follow-up or the time of disease progression or relapse or death from any cause (up to approximately 72 months)
  Progression-free survival (PFS) was defined as the time from randomization to the last follow-up or the time of disease progression or relapse or death from any cause.
The incidences and types of adverse events (AE) and severe adverse events (SAE) | From enrollment to 90-day after the last dose administration (up to approximately 39 months)
  The incidences and severity of adverse events that occur during treatment will be evaluated according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.3

CONTACTS AND LOCATIONS:
Overall Officials: Jiren Yu, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (8):
- China (8):
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - Lishui Central Hospital, Lishui, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - Ningbo Medical Center LiHuiLi Hospital, Ningbo, Zhejiang
  - Ningbo Second Hospital, Ningbo, Zhejiang
  - Taizhou Hospital, Taizhou, Zhejiang